CLINICAL TRIAL: NCT04223011
Title: Initiating Substance Use Disorder Treatment for Hospitalized Alcohol Use Disorder Patients: A Pilot Study of Recovery Coaches
Brief Title: Initiating Substance Use Disorder Treatment for Hospitalized Alcohol Use Disorder Patients
Acronym: ISTAP
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to COVID-19, recruitment was halted before we were able to enroll participants. Currently we are unable to resume recruitment due to study staff changes.
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Joji Suzuki, MD, Director, Division of Addiction Psychiatry, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019P003863; 1K23DA042326-01A1 (NIH)
Record Dates: First submitted 2020-01-07; First posted 2020-01-10 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- In-Hospital Recovery Coach Intervention (Experimental): As this is a single-arm, open-label study, all subjects will receive the interventional arm, specifically in-hospital manualized sessions with the recovery coach.
  Interventions: Behavioral: In-Hospital Recovery Coach Intervention

INTERVENTIONS:
Behavioral: In-Hospital Recovery Coach Intervention — The recovery coach will meet with the patient at least once during the hospital admission, during which he/she will reinforce the importance of continuing medication treatments, if initiated, as well as community and social supports for recovery and will discuss the plan for engaging in these services. This will include recommendations for suitable community resources for recovery services, or for housing, transportation, or other external barriers that may make it more difficult to engage in outpatient treatment. The recovery coach will encourage the participant to complete a relapse prevention plan, and help the patient organize post-discharge appointments and review medications. If applicable, family members and significant others will be encouraged to be present for these encounters.

SUMMARY:
The purpose of this study is to evaluate the impact of a manualized in-hospital recovery coach intervention on rates of post-discharge treatment retention and alcohol use among hospitalized patients with alcohol use disorder.

DETAILED DESCRIPTION:
Patients with alcohol use disorder (AUD) are susceptible to a variety of medical, psychiatric, and social complications, and utilize acute health services frequently; the prevalence of hospitalized patients with AUD is estimate to be between 16% and 26%. While the treatment for the acute complications of AUD such as withdrawal or seizures are treated adequately in the hospital setting, there is a growing recognition that hospitalizations should be utilized as opportunities to initiate treatment for the underlying substance use disorder that likely played a role in the hospitalization in the first place. A large majority (90%) of individuals with active AUD are not engaged with any formal treatment. A promising approach so far in engaging AUD patients has been Screening, Brief Intervention, and Referral to Treatment (SBIRT), particularly for at-risk drinkers (i.e. binge drinkers but not meeting criteria for AUD). However, studies of SBIRT alone is insufficient in reducing alcohol use in heavily dependent, hospitalized patients with alcohol use disorder. Engagement with hospital-based addiction consultation services is helpful with linkage to treatment after discharge, but nearly half of the referred patients never make it to their first appointment. Given the complex medical and psychosocial needs of hospitalized AUD patients, more research on care management interventions that focus on the transitions of care for AUD patients may be needed. There is a growing body of evidence for the benefits of recovery coaches, who provide peer-delivered support services, to help SUD patients in the community. Tracing their origin to mutual support groups to supplement traditional clinical services, recovery coaches are individuals with lived experience of recovery, and are referred to by a variety of names in the literature (i.e. consumer providers, peer support specialists, peer workers, peer mentors). Recovery coaches typically provide services in four domains: 1) emotional (demonstrate empathy, bolster confidence, and foster hope), 2) informational (share knowledge and help skill-building), 3) instrumental (provide assistance with housing, employment, transportation, etc.), and 4) affiliational (create community and sense of belonging). Studies of recovery coaches have demonstrated greater treatment retention, reduced substance use, and reduced inpatient utilization. However, no prior studies have examined the impact of recovery coaches specifically in improving hospitalized AUD patients link with outpatient treatment. As such, the aim of this study is to evaluate the impact of a in-hospital recovery coach intervention on rates of post-discharge treatment retention and alcohol use among hospitalized patients with alcohol use disorder.

ELIGIBILITY:
Inclusion Criteria:

* English speaking, adults aged 18-75
* Diagnosis of DSM-5 alcohol use disorder, severe, actively using alcohol until the time of hospitalization
* Not engaged in SUD treatment including 12-steps within 1 month of hospital admission
* Are being referred to the BWH Bridge Clinic or the BWFH ARP for ongoing SUD treatment after discharge

Exclusion Criteria:

* DSM-5 diagnosis of opioid use disorder
* Unable to provide informed consent due to mental status

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Treatment retention in substance use disorder treatment | 4 weeks following hospitalization discharge date
  Following discharge, the electronic health record of the participant will be examined to confirm whether the participant was successfully seen at the Brigham and Women's Hospital Bridge Clinic or the Brigham and Women's Faulkner Hospital Addiction Recovery Program by checking the visit notes. The proportion of participants who are successfully linked will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Joji Suzuki, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No